CLINICAL TRIAL: NCT00410709
Title: A Phase 1B Single Treatment, Pharmacokinetic and Tolerance Study of NatroVA Topical Creme (1%) i Pediatric Subjects 6 to 24 Months of Age
Brief Title: A Pharmacokinetic (PK) Study of NatrOVA Topical Creme (1%) in Pediatric Subjects 6 to 24 Months of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ParaPRO LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPN-106-06
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2008-08-01 (Estimated); Status verified 2008-07

CONDITIONS: Pediculosis Capitis (Head Lice)
Keywords: Pediculosis Capitis; Head Lice; Crawlers; Ova; Nits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: NatrOVA Creme Rinse (1%)

SUMMARY:
This is an open label, single center, single dose PK study of NatrOVA Creme Rinse (1%), an investigational treatment for head lice and nits, in normal, healthy infants.

DETAILED DESCRIPTION:
There are millions of children and adults affected with head lice each year in the United States. It has become a major nuisance in school children resulting in many lost school days and frustrated parents. Lice and nit resistance to current OTC products is being widely reported. Compliance with product instructions is thought to be low. Therefore a safe and effective alternative to these products is desirable.

Spinosad (the active ingredient in NatrOVA) and its formulations have been approved as agricultural insecticides in the US, Canada and Australia, and has received provisional approval in the UK, Spain and several other European Union countries.

Spinosad is being formulated into a creme rinse product (NatrOVA) using excipients that are widely used and are "generally regarded as safe" (GRAS)

This study is intended to measure the absorption (or lack thereof) of Spinosad through the scalp of infants aged 6 to 24 months, as well as to observe any adverse events related to use of the study drug. A validated method for determining the levels of Spinosad in plasma will be utilized.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 6 to 24 months of age
2. Individuals in good general health, free of any systemic or dermatologic disorders which will interfere with the study results.
3. Completion of an appropriate Informed Consent Agreement.
4. Subjects must be available to stay in the clinic for blood draws. Parents or guardians must be available to stay in the clinic with the minor subject, for the duration of the study.
5. Subjects must have veins capable of withstanding multiple blood draws.
6. Normal values (at screening) for serum chemistry and hematology for subjects.

Exclusion Criteria:

1. History of irritation or sensitivity to pediculicide or hair care products or ingredients.
2. History of known allergy or sensitivity to topical anesthetics including lidocaine and prilocaine.
3. Systemic diseases that could interfere with the results of this study.
4. Any condition or illness that, in the opinion of the Principal Investigator or designee, may compromise the objectivity of the protocol or the safety of the subject.
5. The use of antibiotics or other systemic medications within two weeks of the screening visit, which in the opinion of the investigator, could interfere with the outcome of the study.
6. Participation in a previous drug study within the past 30 days.
7. Individuals with any visible skin/scalp condition at the treatment site which will interfere with the evaluations according to the opinion of the Investigator.
8. Parents or guardians who, in the opinion of the Investigator, do not understand their child's requirements for study participation and/or may be likely to exhibit poor compliance.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2006-12; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Safety: Frequency of Adverse events and scalp evaluations for irritation | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Brown, MD, Principal Investigator — Hill Top Research
Locations (1):
- Hill Top Research, St. Petersburg, Florida, United States